CLINICAL TRIAL: NCT03948464
Title: Repurposing Slow-Release Oral Morphine as a New Oral Alternative for the Treatment of Opioid Use Disorder
Brief Title: Slow-Release Oral Morphine for the Treatment of Opioid Use Disorder
Acronym: pRESTO
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study unable to proceed per protocol due to COVID-19 precautions
Sponsor: M. Eugenia Socias (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Vancouver Foundation (Other); Mayne Pharma International Pty Ltd (Industry)
Responsible Party: Sponsor-Investigator, M. Eugenia Socias, Research Scientist, BC Centre on Substance Use
Organization: BC Centre on Substance Use (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BCCSU-002
Record Dates: First submitted 2019-05-07; First posted 2019-05-14 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Opioid-Related Disorders; Opiate Substitution Treatment; Morphine; Methadone; Fentanyl
Keywords: slow-release oral morphine; methadone; opioid use disorder; fentanyl
MeSH Terms: conditions — Opioid-Related Disorders | interventions — Morphine; Methadone

STUDY DESIGN:
Intervention Model Description: 1:1 randomization
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Slow release oral morphine (SROM) (Experimental): Daily witnessed ingestion of SROM (24-hour formulation) for 24 weeks as per provincial and national guidelines for opioid use disorder.
  Interventions: Drug: Slow release oral morphine (SROM)
- Methadone (Active Comparator): Daily witnessed ingestion of methadone for 24 weeks as per provincial and national guidelines for opioid use disorder.
  Interventions: Drug: Methadone

INTERVENTIONS:
Drug: Slow release oral morphine (SROM) — Slow release oral morphine is an opioid agonist. Slow release oral morphine will be administered via daily witnessed ingestion at designated community pharmacies.
  Other Names: Kadian
  Arms: Slow release oral morphine (SROM)
Drug: Methadone — Methadone is an opioid agonist. Methadone will be administered via daily witnessed ingestion at designated community pharmacies.
  Other Names: Methadose/ Metadol D/Compounded methadone
  Arms: Methadone

SUMMARY:
This is a non-inferiority randomized clinical trial that will compare slow release oral morphine vs methadone as a second line oral treatment for opioid use disorder.

DETAILED DESCRIPTION:
Slow-release oral morphine (SROM) has emerged as a promising yet understudied form of oral treatment for opioid use disorder (OUD), with preliminary studies suggesting similar efficacy rates as methadone with respect to promoting abstinence, and with better improvements in a number of patient-reported outcomes, including tolerability, treatment satisfaction, mental symptoms, and craving. The proposed study is an open-label, non-inferiority, randomized controlled trial evaluating the relative effectiveness, safety and acceptability of SROM vs. methadone for the treatment of OUD in outpatient clinical settings. Participants will be randomized 1:1 to SROM or methadone for 24 weeks. Data linkages performed three years after randomization will evaluate long term health outcomes. This study aims to provide evidence to optimize care for individuals with OUD, and potentially increase access to additional form of evidence-based oral treatment.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all the following criteria to be eligible for the study:

1. Be between 19 and 65 years of age, inclusively;
2. Be diagnosed with opioid use disorder requiring opioid agonist treatment (OAT), as per DSM-5 (Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition) criteria and the discretion of the study physician;
3. Be interested in receiving OAT;
4. Be willing and eligible to be randomized to slow release oral morphine (SROM) or methadone-based OAT as per British Columbia guidelines;
5. If female:

   1. Be of non-childbearing potential, defined as (i) postmenopausal (12 months of spontaneous amenorrhea and over 45 years of age); or (ii) documented surgical sterilization (i.e., tubal ligation, hysterectomy, or bilateral oophorectomy); or
   2. If of childbearing potential, be willing to use an acceptable method of contraception throughout the study and have a negative pregnancy test at screening;
6. Be able to provide written informed consent;
7. Be willing to comply with study procedures;
8. Be able to communicate in English;

Exclusion Criteria:

Participants will be excluded from the study if any of the following criteria are met:

1. Any disabling, severe, or unstable medical or psychiatric condition that, in the opinion of the study physician, precludes safe participation in the study or the ability to provide fully informed consent, as assessed by medical and psychiatric history, physical examination, vital signs, and/or laboratory tests. These may include but are not limited to: significant respiratory depression, severe respiratory compromise or obstructive disease, severe respiratory distress, acute or severe bronchial asthma, known or suspected paralytic ileus;
2. Any severe or unstable co-morbid substance use disorder (e.g., delirium tremens, acute alcohol intoxication) that, in the opinion of the study physician, precludes safe participation in the study;
3. Maintenance on buprenorphine at doses of ≥4 mg in the 5 days prior to screening and stable in the opinion of the study physician;
4. Maintenance on methadone at doses of ≥60 mg in the 5 days prior to screening and stable in the opinion of the study physician;
5. Maintenance on slow release oral morphine at doses of ≥250 mg in the 5 days prior to screening and stable in the opinion of the study physician;
6. Pregnant, breastfeeding, or planning to become pregnant during the study period;
7. History of a serious adverse drug reaction, hypersensitivity reaction, or allergy to methadone or SROM;
8. Use of an investigational drug in the 30 days prior to screening;
9. Pending legal action or other reasons that might prevent completion of the study;
10. Current or anticipated need for treatment with any medication that may interact with methadone or SROM (e.g., benzodiazepines, monoamine oxidase inhibitors [MAOIs] pRESTO Protocol Version 3.0, 08 October 2019 Page 21 of 66 used currently or within the past 14 days) and that, in the opinion of the study physician, would be deemed unsafe or could prevent study completion.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Opioid Use | 24 weeks
  This will be measured by the overall proportion of opioid-free urine drug screens during the 24 weeks of active treatment (excluding the assigned therapy and it's metabolites), with missing samples defined as being positive for opioids

SECONDARY OUTCOMES:
Treatment Retention | 24 weeks
  Treatment retention will be measured by the proportion of participants on the assigned opioid agonist treatment (OAT) at the end of the study, defined as having both a) an active prescription for the assigned OAT at week 24, and b) a positive urine drug screen result for the assigned OAT at week 24.
Adverse Events Related to Study Medications | 24 weeks
  The safety of each study medication will be evaluated by monitoring and gathering information on adverse events (AE) and serious adverse events (SAE), including overdoses, from the time of treatment initiation until the Safety Follow-up Visit. AEs and SAEs will be summarized by MedDRA (Medical Dictionary for Regulatory Activities) System Organ Class and Preferred Term, and the frequency and nature of AEs and SAEs will be compared across treatment arms.
Number of Overdose Events | 24 weeks
  Non-fatal overdoses since the previous visit will be assessed at baseline and every 12 weeks during the 24-week active treatment period, through a combination of self-report and participant's medical record. Data on fatal overdoses will be captured using vital statistics, and supplemented with information from contacts.
Treatment Satisfaction: Medication Satisfaction Questionnaire (MSQ) | 24 weeks
  Participant satisfaction with the assigned treatment will be assessed through administration of the Medication Satisfaction Questionnaire (MSQ) at weeks 4, 12 and 24 of the study. This single-item patient-completed questionnaire evaluates participant's satisfaction with treatment medication on a 7-point Likert scale ranging from "extremely dissatisfied" to "extremely satisfied."
Psychological Functioning | 24 weeks
  Psychological functioning will be measured by the "PROMIS (Patient-Reported Outcomes Measurement Information System) Emotional Distress -Anxiety-Short Form" and the "PROMIS Emotional Distress-Depression-Short Form" measures for anxiety and depression. These instruments will be administered at baseline, as well as at weeks 4, 12 and 24. These measures sum the frequency with which a participant experiences symptoms of depression and anxiety.
Changes in Drug-Related Problems | 24 weeks
  The Addiction Severity Index (ASI) Self-Report Form will be used to assess changes in drug-related problems between baseline and week 24. The ASI has 34 questions. The answer value of each question is divided by its maximum answer value and the total number of questions, and the individual results are then summed to create a composite value.
Changes in Quality of Life: EQ-5D-5L | 24 weeks
  Changes in health-related quality of life (HRQoL) between baseline and the end of treatment will be measured by the EuroQol "EQ-5D-5L" tool. The EQ-5D-5L will be administered at baseline and every 4 weeks during the 24-week active treatment period. The EQ-5D-5L includes a 5-level descriptive system and a visual analogue scale.The descriptive system has five categories (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression), each of which will be rated on a scale of 1 to 5 with 1 being the least severe and 5 being the most severe. The visual analogue scale is a vertical scale from 0 to 100, with 0 labelled "the worst health you can imagine" and 100 labelled "the best health you can imagine."
Opioid Craving | 24 weeks
  Opioid cravings over time will be measured using a 100 mm visual analog scale (VAS). The VAS will be administered at baseline, week 2, week 4, and every 4 weeks for the remainder of the 24-week active treatment period. The VAS is a horizontal scale with 11 lines labeled from left to right with the numbers "0" to "10", and word anchors at each end representing the extremes, where "0=no craving" and "100 mm=most intense craving".
Other Substance Use | 24 weeks
  Use of other substances will be measured using the Timeline Follow-Back (TLFB) instrument, which will be administered at baseline and every study visit thereafter.

CONTACTS AND LOCATIONS:
Overall Officials: M. Eugenia Socias, MD, MSc, Principal Investigator — BC Centre on Substance Use
Locations (1):
- BCCSU Cordova Office, Vancouver, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No